CLINICAL TRIAL: NCT04205630
Title: A Single-arm Phase II Trial to Evaluate the Safety and Efficacy of the Antibody-Drug Conjugate (ADC) SYD985 in Patients With Human Epidermal Growth Factor Receptor 2 (HER2)-Expressing Endometrial Carcinoma Who Previously Progressed on or After First Line Platinum-based Chemotherapy
Brief Title: SYD985 in Patients With HER2-expressing Recurrent, Advanced or Metastatic Endometrial Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Byondis B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYD985.003
Record Dates: First submitted 2019-12-12; First posted 2019-12-19 (Actual); Results first posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — trastuzumab duocarmazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SYD985 (Experimental): SYD985, Intravenous, every 3 weeks (Q3W)
  Interventions: Drug: SYD985

INTERVENTIONS:
Drug: SYD985 — SYD985 powder for concentrate for solution for infusion
  Other Names: Trastuzumab vc-seco-DUBA; (vic-)trastuzumab duocarmazine

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of SYD985 in recurrent, advanced or metastatic endometrial cancer.

DETAILED DESCRIPTION:
This is an open-label, single-arm study in patients with HER2-expressing recurrent, advanced or metastatic endometrial carcinoma. HER2-expression is defined as a 1+, 2+ or 3+ score on immunohistochemistry (IHC) or positive by in situ hybridization (ISH). Eligible patients for this study should have progressed on or after first line platinum-based chemotherapy. Patients who have had two or more lines of chemotherapy for advanced/metastatic disease are not eligible.

Eligible patients will receive SYD985 until disease progression or unacceptable toxicity. Patients who have stopped study treatment for other reasons than disease progression will continue their tumor evaluations in an observation period until disease progression or start of a new anticancer therapy.

ELIGIBILITY:
Main Inclusion Criteria:

* Females with histologically confirmed recurrent, advanced or metastatic endometrial carcinoma
* Eligible patients should have progressed on or after first line platinum-based chemotherapy for advanced/metastatic endometrial cancer. Patients who have had two or more lines of chemotherapy for advanced/metastatic disease are not eligible, taking into account the following:

  * Patients may have received up to one additional line of chemotherapy if given in the neoadjuvant or adjuvant setting. If such treatment was completed less than 6 months prior to the current tumor recurrence or progression it is to be considered first-line treatment;
  * No more than one line of non-cytotoxic systemic cancer therapy (such as immunotherapy, trastuzumab or protein kinase inhibitors) is allowed.
* HER2 tumor expression defined as a 1+, 2+ or 3+ score on IHC or positive by ISH
* At least one measurable cancer lesion as defined by the Response Evaluation Criteria for Solid Tumours (RECIST version 1.1);
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2;

Exclusion Criteria:

* Current or previous use of a prohibited medication as listed in the protocol;
* History of infusion-related reactions and/or hypersensitivity to trastuzumab;
* History of keratitis;
* Severe, uncontrolled systemic disease at screening;
* Left Ventricular Ejection Fraction (LVEF) < 50%, or a history of clinically significant decrease in LVEF during previous treatment with trastuzumab;
* History of clinically significant cardiovascular disease;
* Symptomatic brain metastases, brain metastases requiring steroids to manage symptoms, or treatment for brain metastases within 8 weeks prior to randomization;
* History or presence of idiopathic pulmonary fibrosis, organizing pneumonia (e.g. bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Byondis B.V., The Netherlands
Locations (36):
- Smilow Cancer Hospital (Yale), New Haven, Connecticut, United States
- Poland (2):
  - MedTrials, Krakow
  - St. John of Dukla Oncology Center of Lublin Land, Lublin
- Russia (12):
  - Arkhangelsk Clinical Oncology Center, Arkhangelsk
  - Chelyabinsk Regional Clinical Oncology and Nuclear Medicine Center, Chelyabinsk
  - Regional Oncology Center, Irkutsk
  - Clinical Oncology Center, Omsk
  - Orenburg Regional Clinical Oncology Center, Orenburg
  - Oncology Center of Moskovskiy District, Saint Petersburg
  - Private Medical Institution "EVROMEDSERVIS", Saint Petersburg
  - AV Medical Group, Saint Petersburg
  - Oncology Center #2, Sochi
  - Tambov Regional Oncological Clinical Center, Tambov
  - Republican Clinical Oncology Center, Ufa
  - Volgograd Regional Clinical Oncology Center, Volgograd
- Serbia (3):
  - National Cancer Research Center, Belgrade
  - Oncology Institute of Vojvodina (IOV), Clinic of Surgical Oncology, Department of Gynecology, Kamenitz
  - Clinical Center Nis, Clinic of Oncology, Niš
- Singapore (2):
  - National University Hospital, Department of Hematology-Oncology, Singapore
  - National Cancer Centre Singapore, Singapore
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Ukraine (11):
  - Cherkasy Regional Oncology Dispensary of Cherkasy Oblast Council, Cherkasy
  - Chernivtsi Regional Clinical Oncology Center, Chernivtsi
  - "City Clinical Hospital #4" under Dnipro City Council, Dnipro
  - Prykarpattia Clinical Oncology Center, Ivano-Frankivsk
  - State Institution: S.P. Hryhoriev Institute of Medical Radiology under the Ukrainian Academy of Medical Sciences, Kharkiv
  - Communal Non-profit enterprise "Regional Center of Oncology", Kharkiv
  - Medical Center "Verum", Kyiv
  - Odesa Regional Clinical Hospital, Odesa
  - Public Non-Profit Enterprise Ternopil Regional Clinical Oncology Center, Ternopil
  - Podilla Regional Oncology Center, Vinnytsia
  - Medical Center ONCOLIFE LLC, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 80 participants were screened, out of which 64 patients were enrolled in the study.
Groups:
- SYD985: SYD985, Intravenous, 1.2 mg/kg once every 3 weeks (Q3W)
Period: Overall Study
Arm/Group | SYD985
Started | 64
Full Analysis Set (All Patients Who Received at Least 1 Dose of Study Treatment) | 64
Efficacy Analysis Set (All Patients Who Had at Least One Post-baseline Tumour Evaluation Assessment) | 61
Completed | 0
Not Completed | 64
Not completed — Disease progression per RECIST 1.1 | 37
Not completed — Disease clinical progression | 7
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 17
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Groups:
- SYD985: SYD985, Intravenous, every 3 weeks (Q3W)
  SYD985: Powder for concentrate for solution for infusion
Arm/Group | SYD985
Number analyzed (Participants) | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (7.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 64
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 13
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 48
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 7
  Singapore | 5
  United States | 9
  Ukraine | 19
  Poland | 4
  Serbia | 6
  Russia | 14

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the proportion of patients with an assessed best overall response of complete response or partial response according to Response Evaluation Criteria In Solid Tumors (RECIST) v1.1.
Time Frame: 2 years
Population: Efficacy analysis set (EAS) was used for the efficacy analyses. The EAS consists of a subset of the full analysis set (FAS) patients who had a baseline and at least one post-baseline tumour evaluation assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | SYD985
Number analyzed (Participants) | 61
Participants | 20

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from the date of randomization to the date of first documented disease progression by investigator assessment according to RECIST v1.1 or death due to any cause, whichever occurred earlier.
Time Frame: 2 years
Population: Progression-free survival is measured for the Full Analysis Set (FAS).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SYD985
Number analyzed (Participants) | 64
months | 5.6 [4.0 to 7.6]

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from date of randomization to death due to any cause.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SYD985
Number analyzed (Participants) | 64
months | 16.3 [11.6 to 20.5]

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs)
Description: AEs will be graded by the investigator as assessed by CTCAE v5.0.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | SYD985
Number analyzed (Participants) | 64
Participants | 51

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each participant from the time of signing the main informed consent form (ICF) up to 30 days after the treatment discontinuation visit, up to 2 years 9 months.
Arm/Group | SYD985
All-Cause Mortality (participants affected / at risk) | 36/64
Serious Adverse Events (participants affected / at risk) | 12/64
Other Adverse Events (participants affected / at risk) | 51/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SYD985 (N=64)
Abdominal hernia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 1
COVID-19 pneumonia (Infections and infestations) | 3
Anaemia (Blood and lymphatic system disorders) | 2
Cardiac failure (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
General physical health deterioration (General disorders) | 1
Sudden death (General disorders) | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SYD985 (N=64)
Keratitis (Eye disorders) | 20
Dry eye (Eye disorders) | 18
Conjunctivitis (Eye disorders) | 14
Periorbital oedema (Eye disorders) | 7
Lacrimation increased (Eye disorders) | 5
Vision blurred (Eye disorders) | 5
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 11
Alopecia (Skin and subcutaneous tissue disorders) | 7
Fatigue (General disorders) | 9
Pyrexia (General disorders) | 6
Anaemia (Blood and lymphatic system disorders) | 8
Leukopenia (Blood and lymphatic system disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Nausea (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 4
Dry mouth (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 4
Dysgeusia (Nervous system disorders) | 5
Peripheral sensory neuropathy (Nervous system disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 7
Infusion related reaction (Injury, poisoning and procedural complications) | 8
Weight decreased (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agrees to provide to the Sponsor 60 days prior to intended submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the study. The Sponsor has the right to review and comment with respect to publications, abstracts, slides, and manuscripts including the data analysis and presentation. In case of disagreement, efforts will be undertaken to resolve any such issues, but the ultimate decision remains with the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/30/NCT04205630/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-19): https://cdn.clinicaltrials.gov/large-docs/30/NCT04205630/SAP_001.pdf